CLINICAL TRIAL: NCT02429362
Title: Obstetrical Repository of Biological Materials
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Collaborators: Regional One Health (Other); University of Tennessee Regional One Physicians (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14-03383-XP
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Health Problems in Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Sample collections for purposes of: understanding of normal events in pregnancy; disease conditions of the woman/baby during pregnancy; and future use in studies to develop cell lines for research, create tests to diagnose disease, or develop treatments.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women & their stillborn infants: All English speaking female patients who are seen in the Regional One Health perinatal clinics and/or deliver at Regional One Health are the group of study's focus. Likewise, when a delivery results in a stillbirth, the stillborn baby will also be an additional group of our study's focus.

SUMMARY:
Subjects are being asked to donate blood, urine, vaginal secretions and/or tissue to a repository for research.This repository will store donated specimens for future research. The Department of Obstetrics and Gynecology at the University of Tennessee Health Science Center, under the direction of Dr. Giancarlo Mari, Professor and Chair, is responsible for the operation of the repository.

Additionally, in the case of a stillborn child, the mother will be given the opportunity to donate samples from her stillborn baby's autopsy to a repository for research.

DETAILED DESCRIPTION:
The stored samples will be used in studies to help researchers understand normal events in pregnancy, as well as events that occur when women and/or their babies have a disease or condition during pregnancy. Additionally, the samples may be used in future studies to develop cell lines for research, create tests to diagnose disease, or develop treatments. A cell line is the result of cells grown outside the body in a laboratory. This process will allow those cells to grow continuously when given the appropriate nutrients and conditions for growth, and will result in a permanent cell culture which is the collection of cells that are grown outside the body in a laboratory.

The stored samples will also be used in future studies to help researchers identify genetic influences during pregnancy. Genes are like blueprints in each of your cells that determine traits that you inherit, like eye color and hair color. Genes may also influence what diseases you get and how you respond to treatment. DNA is the substance that makes up your genes.

The subject will sign an informed consent for her participation (Primary Informed Consent). In the situation of a stillbirth occurring, the mother of the stillborn baby will sign an informed consent regarding the tissue samples to be obtained during the hospital's routinely performed autopsy. (Secondary Informed Consent).

ELIGIBILITY:
Inclusion Criteria:

* English speaking female
* patients presenting for medical care at the Regional One Health perinatal clinics or Regional One Health Labor and Delivery Dept. will be asked to participate in the study.

Exclusion Criteria:

* Those not meeting the above criteria.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All English speaking female patients who are seen in the Regional One Health perinatal clinics and/or deliver at Regional One Health will be asked to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Maternal biological sample collection for repository | On average, samples will be collected up to 42 wks of pregnancy & also at time of delivery.
  Outcomes will be assessed (including morbidity and mortality associated with the pregnancy/delivery). Studies of specimens may involve examinations for gross pathology, infection, or genomic/proteomic/metabolomic analyses.

SECONDARY OUTCOMES:
Stillborn fetal sample collection for repository | At the occurence of a stillbirth, study samples will be collected from the stillborn baby following the hospital's stillborn autopsy policy, on average by the end of 1 week post delivery.
  Outcomes will be assessed (including morbidity and mortality associated with the pregnancy/delivery). Studies of specimens may involve examinations for gross pathology, infection, or genomic/proteomic/metabolomic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Mari, M.D., Principal Investigator — Prof. & Chair, UTHSC; Dir.,TN Inst. of Feto-Maternal & Infant Health; Dir., High-Risk Obstetrics Ctr of Excell., Regional Medical Ctr
Locations (1):
- University of Tennessee Health Science Center, OB-GYN, Memphis, Tennessee, United States